CLINICAL TRIAL: NCT04326699
Title: Therapeutic Potentials of Bilateral Sacroiliac Joint Injection in Lumbar Disc Prolapse: a Prospective Study
Brief Title: Bilateral Sacroiliac Joint (SIJ) Injection in Lumbar Disc Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Associate professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 15/3/2020
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Lumbar Disc Herniation; Sciatica; Low Back Pain, Mechanical; Spine Stiffness
Keywords: Disc Prolapse; sacroiliac joint; Injection; Ultrasound
MeSH Terms: conditions — Intervertebral Disc Displacement; Sciatica; Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacroiliac joint injection group (Active Comparator): The active group will receive bilateral sacroiliac joint injection of 1 mL 2 % lidocaine hydrochloride (xylocaine, AstraZeneca) mixed with triamcinolone 40 milligrams (Kenacort, Bristol Myers Squip) under ultrasound guidance.
  Interventions: Procedure: Bilateral SIJ injection
- control group (No Intervention): The other group will not receive the sacroiliac joint injection

INTERVENTIONS:
Procedure: Bilateral SIJ injection — under US guidance a 22G spinal needle, where 1 mL 2 % lidocaine hydrochloride (xylocaine, AstraZeneca) mixed with triamcinolone 40 milligrams (Kenacort, Bristol Myers Squip) will be injected in each SIJ
  Arms: Sacroiliac joint injection group

SUMMARY:
Bilateral sacroiliac joint injection in symptomatic lumbar disc prolapse under ultrasound guidance and studying the effect of this technique on pain, spine mobility and activity of daily living.

DETAILED DESCRIPTION:
86 Patients with lumbar disc prolapse diagnosed by either MRI or CT will be included. All of them aged > 18 years with no special condition for the duration of disc prolapse. All of them had clinical manifestations in the form of mechanical low back pain or sciatica or limited spine mobility. All participants had no or poor response to conservative treatment. Previous surgery, severe facet arthropathy, ankylosing spondylitis, sensory or motor deficit and wedge fracture were considered as exclusion criteria. Distraction, compression, thigh thrust, and sacral thrust were used to assess SIJ dysfunction only at baseline before injection. Fingertip to floor and Oswestry disability index (ODI) were used to assess mobility and function of the spine at baseline (before and after injection) and after 2 and 16 weeks. Visual Analogue Scale (VAS) was used for pain appraisal at the same intervals. Participants will be randomly assigned into active and control group using 1:1 allocation. In the active group bilateral SIJ injection will be performed under ultrasound US guidance. Under US guidance a 22G spinal needle, where 1 mL 2 % lidocaine hydrochloride (xylocaine, AstraZeneca) mixed with triamcinolone 40 milligrams (Kenacort, Bristol Myers Squip) will be injected in each SIJ.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar disc prolapse diagnosed by either MRI or CT were included.
* All of them aged > 18 years
* No special condition for the duration of disc prolapse.
* All of them had clinical manifestations in the form of mechanical low back pain or sciatica or limited spine mobility.
* All participants had no or poor response to conservative treatment

Exclusion Criteria:

* Previous surgery
* Severe facet arthropathy
* Ankylosing spondylitis
* Sensory or motor deficit
* Wedge fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Pain assessment by visual analogue scale. | at baseline 0 time, after 2 weeks and after 16 weeks
  Visual analogue scale, 0 means no pain and 10 means the maximum possible pain.
Spine mobility, finger tip to floor test | Baseline 0 time, after 2 weeks and after 16 weeks
  comparison to the intial values with each visit to detect changes with no definite references.
Oswestry disability index | Baseline 0 time, after 2 weeks and after 16 weeks
  0 value means no disability and 100 means complete disability

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt